CLINICAL TRIAL: NCT07220330
Title: An Investigational Study Examining the Cross-Validation of QbMobile in ADHD and Normative Populations
Status: Enrolling by invitation | Type: Observational
Sponsor: Qbtech AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 00082479 / QB24-01
Record Dates: First submitted 2025-10-15; First posted 2025-10-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: No History of ADHD; Attention Deficit Hyperactivity Disorder (ADHD); Healthy Volunteer
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This single cohort includes subjects with and without ADHD.: Eligible participants that do not have a documented or suspected current or lifetime diagnosis of ADHD will be recruited from the general population using different recruitment activities (letters, posted flyers, etc.).
  Eligible participants being referred for their initial assessment or have a diagnosis of ADHD but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: QbMobile

INTERVENTIONS:
Device: QbMobile — QbMobile is a software application that can be installed on a smartphone device used to measure activity, attention, impulsivity, and movement patterns in participants over a two-day period.

SUMMARY:
The purpose of this study is to investigate QbMobile ability to collect and provide accurate and objective data which can be used to facilitate assessment and treatment procedures for ADHD in a clinical setting as well as remotely.

DETAILED DESCRIPTION:
This study aims to evaluate the performance of QbMobile in children, adolescents, and adults from the normative population, those referred for an initial ADHD assessment, and individuals with an ADHD diagnosis who are not currently receiving ADHD treatment.

Participants will complete the 10-minute QbMobile test on their personal device during a scheduled clinical visit. They will then repeat the test remotely the following day at the same time as the previous test +/-3 hours.

For participants referred for an ADHD assessment or a has an ADHD diagnosis, QbMobile must be completed prior to initiating any ADHD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (including parent/legal guardians consent when this is required for individuals under 18 years old and assent as is required based on the age of participant) for QbMobile;
* Aged > 6 years and < 60 years old;
* Have no documented or suspected current or lifetime diagnosis of ADHD or referred for an initial assessment for ADHD or have a diagnosis of ADHD but not currently receiving treatment;
* Meet DSM-5 or ICD-11 criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactivity/impulsive presentation) per sites standard clinical care evaluation;
* Qbtech Rating Scale total score of >24 at Visit 1;
* Have adequate sensory and physical ability to complete QbMobile;
* Possess or has access to an iPhone model that supports QbMobile.

Exclusion Criteria:

* Intellectual disability designated by IQ<75;
* Has used psychostimulant medication within the past 7 days prior to Visit 1;
* A current medical diagnosis that could significantly affect test performance (brain injuries, Parkinson's disease, current epilepsy or active seizures, amyotrophic lateral sclerosis (ALS), multiple sclerosis, dementias (e.g., vascular dementia, Alzheimer disease, etc.);
* Other conditions that could affect test performance (migraine or other types of severe headache, chronic or acute pain);
* Substance use (e.g., alcohol, drugs) that may affect performance on the day of the tests.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Potential study participants who meet the eligibility criteria will be identified through referrals and recruitment efforts at the participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Standardized QbMobile Scores of the four parameters: Attention, Impulsivity, Activity, and Movement Patterns. | 10-minute testing period
  QbMobile generates standardized scores (SD-scores) for attention, impulsivity, activity, and movement patterns using age and sex at birth adjusted norms. These scores provide objective data collected during the 10-minute test session and are automatically included in a standardized report generated immediately upon test completion. This supports evaluation of test validity for ADHD-related symptom measurement.

SECONDARY OUTCOMES:
QbMobile ADHD Symptom Likelihood Score Across Diagnostic Groups | 10 minute testing period
  QbMobile Total score (0-100 where 0 indicates a low likelihood of exhibiting ADHD symptoms and 100 indicates a high likelihood of exhibiting ADHD symptoms) will be compared across participants assessed for ADHD, diagnosed but untreated, and normative participants to evaluate differentiation in ADHD symptom likelihood. This score is automatically generated in the QbMobile report upon test completion.
Comparison of QbMobile SD-Scores Across Testing Environments | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2)
  SD-scores for attention, impulsivity, activity, and movement patterns will be compared between in-clinic and remote QbMobile tests to assess consistency and reliability.
Exploratory Identification of Novel QbMobile Derived Parameters Reflecting Activity, Movement, Attention, and Impulsivity | QbMobile completed at Visit 1 (Day 1) and Visit 2 (Day 2).
  Exploratory analyses will be conducted on raw QbMobile data collected at Visit 1 and Visit 2 to identify potential additional parameters that may serve as indices of activity, attention, impulsivity, and movement. These parameters will be evaluated for their potential association with ADHD symptomatology.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Prodigy Psychiatric Group, San Jose, California
  - Bokhari Medical Consortium, Largo, Florida
  - Nona Pediatric Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the research, limited access to supporting data may be granted upon reasonable request under confidentiality agreements from the corresponding sponsor.